CLINICAL TRIAL: NCT00803803
Title: Dose, Effects and Characteristics of Pilocarpine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Marlene Moster, MD, Attending Surgeon, Wills Eye
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 08-914E
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Open-angle Glaucoma
Keywords: Pilocarpine; POAG; IOP; Concentration; Frequency; Primary open-angle glaucoma; Primary open-angle glaucoma suspect
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilocarpine Concentration (Experimental): Varying concentration 0.5 to 8% - 22 patients were examined regarding: visual acuity, iris color, pupil size, chamber angle, C/D ratio, visual field (VF), coefficient of aqueous outflow and Goldmann tonometry. After a one month washout period, pilocarpine was used 4 times daily, in concentrations from 0.5 to 8%. The amount of IOP change was compared with various clinical findings
  Interventions: Drug: Pilocarpine Concentration
- Pilocarpine Frequency (Experimental): Varying frequency, once to four times daily - 15 patients were included in a crossover study: IOP was checked daily for 3 days and for 9 hours on fourth day. Pilocarpine was started on day 5 once daily OD and BID OS; on day 9 once daily OD and QID OS; on day 12 QID OD and once daily OS; on day 16 once daily OD and QID OS; and on day 19 QID OD and once daily OS. No medications were used on days 23-25. IOP was measured on days 4, 8, 11, 15, 18, 22 and 25.
  Interventions: Drug: Pilocarpine Frequency

INTERVENTIONS:
Drug: Pilocarpine Concentration — Varying concentration 0.5 to 8%
  Arms: Pilocarpine Concentration
Drug: Pilocarpine Frequency — 1 to 4 times daily
  Arms: Pilocarpine Frequency

SUMMARY:
The purpose of this investigation, in which pilocarpine was given in repeated doses, was to evaluate: Part I - the effects of different concentrations of pilocarpine hydrochloride on intraocular pressure. Part II -the effects on intraocular pressure of glaucomatous patients to pilocarpine 2% when given once, twice and four daily. In addition, we studied various attributes of the eye which may serve as indicators of responsiveness of individual patients to pilocarpine.

DETAILED DESCRIPTION:
In addition, we studied various attributes of the eye which may serve as indicators of responsiveness of individual patients to pilocarpine.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma
* Primary open-angle glaucoma suspect

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 1978-08; Primary Completion 1979-08 (Actual); Study Completion 1979-12 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: George L Spaeth, MD, Principal Investigator — Wills Eye Glaucoma Service
Locations (1):
- Wills Eye Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No